CLINICAL TRIAL: NCT00747617
Title: Theca Cell Function in Women With Polycystic Ovary Syndrome
Brief Title: Theca Cell Function in Women With Polycystic Ovary Syndrome (PCOS)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Jeffrey Chang, MD, Principal investigator, University of California, San Diego
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 060679
Record Dates: First submitted 2008-09-04; First posted 2008-09-05 (Estimated); Results first posted 2013-01-29 (Estimated); Last update posted 2018-11-21 (Actual); Status verified 2018-10

CONDITIONS: Polycystic Ovary Syndrome
Keywords: polycystic ovary syndrome; androgens; ovary; LH
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Chorionic Gonadotropin; Ovidrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PCOS group (Active Comparator): Each subject will receive a dose (1, 10, 25, 100, or 250 micrograms) of recombinant human chorionic gonadotropin administered iv on 5 separate occasions.
  Interventions: Drug: recombinant human chorionic gonadotropin
- Control group (Active Comparator): Each subject will receive a dose (1, 10, 25, 100, or 250 micrograms) of recombinant human chorionic gonadotropin administered iv on 5 separate occasions.
  Interventions: Drug: recombinant human chorionic gonadotropin

INTERVENTIONS:
Drug: recombinant human chorionic gonadotropin — Each subject will receive a dose (1, 10, 25, 100, or 250 micrograms) of human chorionic gonadotropin administered intravenously on 5 separate occasions.
  Other Names: Ovidrel

SUMMARY:
The mechanism for increased androgen production in women with polycystic ovary syndrome (PCOS) is not well understood. Excess androgen production by the ovary is stimulated by increased pituitary luteinizing hormone (LH) secretion in this disorder. The investigators hypothesize that in PCOS women ovarian theca cells, which are responsible for androgen synthesis, are more sensitive to LH stimulation compared to that of theca cells from normal women. To test this hypothesis, the investigators propose to conduct a dose-response study in which androgen responses to multiple doses of human chorionic gonadotgropin (hCG), an LH surrogate, will be assessed in PCOS and normal women.

DETAILED DESCRIPTION:
Each subject (normal and PCOS women) will be admitted to the UCSD General Clinical Research Center (GCRC) for study on 5 occasions. All subjects will receive an intravenous injection of hCG dose of 1, 10, 25, 100, and 250 micrograms, each of which will be given on one of 5 different days each separated by at least two weeks at 8 AM. Blood samples will be obtained at t -0.5, 0, and 24 hours after injection. All visits to the GCRC will be done as out patients. The total amount of blood withdrawn will be about 35 teaspoons. For normal control subjects this will be over a period of about 4-6 months and for PCOS subjects this will be over a period of about 6-10 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Normal CBC (Hemoglobin must be at least 11mg/dl)
* Normal renal and liver function tests
* Normal vital signs including normal blood pressure

Exclusion Criteria:

* No oral contraceptives
* No insulin lowering drugs
* No anti-androgens (i.e., spironolactone, flutamide, finasteride, etc)
* No medications that will influence androgen metabolism or clearance
* No medications that will inhibit the cytochrome P450 enzyme system (cimetidine, ketoconozole, etc)
* No use of clomiphene citrate within 3 months prior to study

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2007-09; Primary Completion 2010-04 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: R, Jeffrey Chang, M.D., Principal Investigator — UCSD SChool of Medicine
Locations (1):
- University of California, San Diego, School of Medicine, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chang RJ. The reproductive phenotype in polycystic ovary syndrome. Nat Clin Pract Endocrinol Metab. 2007 Oct;3(10):688-95. doi: 10.1038/ncpendmet0637. PMID 17893687
- [Background] Wachs DS, Coffler MS, Malcom PJ, Shimasaki S, Chang RJ. Increased androgen response to follicle-stimulating hormone administration in women with polycystic ovary syndrome. J Clin Endocrinol Metab. 2008 May;93(5):1827-33. doi: 10.1210/jc.2007-2664. Epub 2008 Feb 19. PMID 18285408
- [Background] Wachs DS, Coffler MS, Malcom PJ, Chang RJ. Comparison of follicle-stimulating-hormone-stimulated dimeric inhibin and estradiol responses as indicators of granulosa cell function in polycystic ovary syndrome and normal women. J Clin Endocrinol Metab. 2006 Aug;91(8):2920-5. doi: 10.1210/jc.2006-0442. Epub 2006 May 23. PMID 16720653
- [Background] Mehta RV, Malcom PJ, Chang RJ. The effect of androgen blockade on granulosa cell estradiol production after follicle-stimulating hormone stimulation in women with polycystic ovary syndrome. J Clin Endocrinol Metab. 2006 Sep;91(9):3503-6. doi: 10.1210/jc.2006-0752. Epub 2006 Jun 27. PMID 16804036
- [Background] Mehta RV, Patel KS, Coffler MS, Dahan MH, Yoo RY, Archer JS, Malcom PJ, Chang RJ. Luteinizing hormone secretion is not influenced by insulin infusion in women with polycystic ovary syndrome despite improved insulin sensitivity during pioglitazone treatment. J Clin Endocrinol Metab. 2005 Apr;90(4):2136-41. doi: 10.1210/jc.2004-1040. Epub 2005 Jan 11. PMID 15644405
- [Background] Chang RJ. A practical approach to the diagnosis of polycystic ovary syndrome. Am J Obstet Gynecol. 2004 Sep;191(3):713-7. doi: 10.1016/j.ajog.2004.04.045. PMID 15467530
- [Derived] Maas KH, Chuan S, Harrison E, Cook-Andersen H, Duleba AJ, Chang RJ. Androgen responses to adrenocorticotropic hormone infusion among individual women with polycystic ovary syndrome. Fertil Steril. 2016 Oct;106(5):1252-1257. doi: 10.1016/j.fertnstert.2016.06.039. Epub 2016 Jul 26. PMID 27473350
- [Derived] Maas KH, Chuan SS, Cook-Andersen H, Su HI, Duleba A, Chang RJ. Relationship between 17-hydroxyprogesterone responses to human chorionic gonadotropin and markers of ovarian follicle morphology in women with polycystic ovary syndrome. J Clin Endocrinol Metab. 2015 Jan;100(1):293-300. doi: 10.1210/jc.2014-2956. PMID 25313914
- [Derived] Cook-Andersen H, Chuan SS, Maas K, Rosencrantz MA, Su HI, Lawson M, Mason HD, Chang RJ. Lack of Serum anti-Mullerian hormone responses after recombinant human chorionic gonadotropin stimulation in women with polycystic ovary syndrome. J Clin Endocrinol Metab. 2015 Jan;100(1):251-7. doi: 10.1210/jc.2014-2948. PMID 25303490
- [Derived] Shayya RF, Rosencrantz MA, Chuan SS, Cook-Andersen H, Roudebush WE, Irene Su H, Shimasaki S, Chang RJ. Decreased inhibin B responses following recombinant human chorionic gonadotropin administration in normal women and women with polycystic ovary syndrome. Fertil Steril. 2014 Jan;101(1):275-9. doi: 10.1016/j.fertnstert.2013.09.037. Epub 2013 Nov 1. PMID 24188875
- [Derived] Rosencrantz MA, Coffler MS, Haggan A, Duke KB, Donohue MC, Shayya RF, Su HI, Chang RJ. Clinical evidence for predominance of delta-5 steroid production in women with polycystic ovary syndrome. J Clin Endocrinol Metab. 2011 Apr;96(4):1106-13. doi: 10.1210/jc.2010-2200. Epub 2011 Jan 26. PMID 21270326

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects recruited from UCSD clinics and coal advertising beginning in 2009 and ending in 2010
Pre-assignment Details: Subjects involved women with PCOS and normal control women undergoing hCG stimulation
Groups:
- PCOS; Normal: Each subject will receive a dose (1, 10, 25, 100, or 250 micrograms) of hCG administered intravenously on 5 separate occasions.
Period: Overall Study
Arm/Group | PCOS | Normal
Started | 13 | 12
Completed | 10 | 11
Not Completed | 3 | 1
Not completed — Lost to Follow-up | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PCOS | Normal | Total
Number analyzed (Participants) | 13 | 12 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 12 | 25
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.5 (1.1) | 30 (1.3) | 29 (1.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 12 | 25
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 13 | 12 | 25

OUTCOME MEASURES:

1. Primary Outcome: Serum 17OHP Responses to hCG
Description: Assess serum 17OHP levels following each dose of hCG adminstration in PCOS and normal subjects
Time Frame: 24 hrs post dose
Population: PCOS and Normal groups were analyzed according to peak 17OHP levels at each dose of r-hCG.
Measure: Mean (Standard Error); unit: ng/ml
Groups:
- PCOS; Normal: Each subject received a dose (1, 10, 25, 100, or 250 micrograms) of iv hCG.
Arm/Group | PCOS | Normal
Number analyzed (Participants) | 10 | 11
ng/ml
  17OHP post 10 micrograms | 2.0 (0.3) | 1.2 (0.1)
  17OHP level post 1 micrograms | 1.1 (0.1) | 1.0 (0.1)
  17OHP level post 25 micrograms | 2.7 (0.3) | 1.7 (0.2)
  17OHP level post 100 micrograms | 3.3 (0.6) | 2.2 (0.3)
  17OHP level post 250 micrograms | 4.0 (0.6) | 2.1 (0.4)
Statistical Analysis 1: Comparison: PCOS vs Normal; Test type: Superiority or Other; p < 0.05, Mixed Models Analysis

2. Secondary Outcome: Serum Testosterone Responses to hCG
Description: Mean serum testosterone levels before and after hCG injection. Serum testosterone levels before (-0.5 and 0 hrs) were averaged to achieve a single value
Time Frame: -0.5, 0, 24 hrs
Measure: Mean (Standard Error); unit: ng/ml
Arm/Group | PCOS | Normal
Number analyzed (Participants) | 10 | 11
ng/ml | 0.6 (0.1) | 0.3 (0.05)

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | PCOS | Normal
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/12
Other Adverse Events (participants affected / at risk) | 0/13 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No